CLINICAL TRIAL: NCT06016868
Title: Identification of a MOLecuLar Signature Predicting Radiosensitivity in Locally Advanced Cervical Cancer Patients (LACC) Treated With Exclusive radiochemotherapY: a Pilot Study
Brief Title: Identification of a MOLecuLar Signature in Locally Advanced Cervical Cancer Patients
Acronym: MOLLY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5773
Record Dates: First submitted 2023-07-25; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional
  Interventions: Procedure: Tumor tissue; Procedure: Blood sample

INTERVENTIONS:
Procedure: Tumor tissue — Each newly diagnosed patient with LACC who meets the inclusion criteria will undergo cervical cancer biopsy either during the outpatient clinical examination or during examination during anesthetic. Part of the biopsy will be sent for histopathological analysis, while the remaining tissue will be embedded in OCT compound and immediately frozen at -80°C prior to transfer to biobank for subsequent analysis.
Procedure: Blood sample — Every patient will undergo a peripheral venous blood sample which will be processed to analyze the presence of the proteins codified by three RNA species (ANXA2-NDRG1-STAT1). This blood sample will be performed before starting the treatment with exclusive CTRT.

SUMMARY:
The importance of radioresistance in cervical cancer treatment failure indicates that certain biomarkers may be useful for cervical cancer treatment individualization. However, to date, no study has analyzed the role of the gene expression signature of the three RNA species (ANXA2-NDRG1-STAT1) to predict radiosensitivity/resistance in cervical cancer patients undergoing exclusive CTRT. The previously validated three-gene signature may enable stratification in LACC patients treated with the current standard of care, represented by exclusive CTRT.

DETAILED DESCRIPTION:
The importance of radioresistance in cervical cancer treatment failure indicates that certain biomarkers may be useful for cervical cancer treatment individualization. Several biomarkers of cervical cancer radioresistance have been previously studied and proposed; however, none of these has been the subject to further clinical studies and implemented into clinical practice. Recently, a panel of three protein coding genes (ANXA2-NDRG1-STAT1) differently expressed in radiosensitive LACC patients compared with the radioresistant ones, has been proposed by our institution. The population of LACC patients included in a previous study was treated with neo-adjuvant CTRT followed by radical surgery. However, to date, no study has analyzed the role of the gene expression signature of the three RNA species (ANXA2-NDRG1-STAT1) to predict radiosensitivity/resistance in cervical cancer patients undergoing exclusive CTRT. The previously validated three-gene signature may enable stratification in LACC patients treated with the current standard of care, represented by exclusive CTRT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix
* FIGO 2018 stage IIB and IIIC1[38]
* Treatment with exclusive chemoradiation including brachytherapy
* Has not previously received any definitive surgical, radiation, or systemic therapy for cervical cancer
* Has radiographically evaluable disease, measurable per RECIST 1.1
* Negative pregnancy test
* Adequate hematologic, renal, and hepatic functions, with following blood tests:

Neutrophils > 1500/μL Platelets > 100.000/ μL Hemoglobin > 9 g/dL Serum creatinine < 1.8 mg/dL Total bilirubin < 3 mg/ dL LDH < 3x normal value GOT < 3x normal value GPT < 3x normal value ALP < 3 x normal value

Exclusion Criteria:

* Rare cervical cancer histologies (neuroendocrine, glassy cells, serous, endometrioid etc)
* Neo-adjuvant treatment
* Patients included in other clinical trials
* Patients refusing to sign informed consent
* Contraindications to radiotherapy
* Contraindications to pelvic radiotherapy: ulcerative colitis, diverticulitis, chronic pelvic inflammatory disease, previous pelvic radiotherapy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix FIGO stage IIB and IIIC1.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
To test the performance of the molecular signature. | 60 months
  To test the performance of the molecular signature in predicting response to exclusive CTRT in LACC patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No